CLINICAL TRIAL: NCT03276429
Title: Development of an Electronic Data Base for Lung Cancer Registry Which Will Include All the Epidemiological, Clinical, Pathological, Molecular and Treatment Parameters in Lung Cancer Patients Who Are Referred to a Tertiary Oncology Unit
Brief Title: Lung Cancer Registry for Lung Cancer Patients
Acronym: LCR
Status: Completed | Type: Observational
Sponsor: Oncology Center of Biochemical Education And Research (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-9MT
Record Dates: First submitted 2017-08-23; First posted 2017-09-08 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Lung Cancer
Keywords: NSCLC; SCLC; MOLECULAR BIOMARKERS
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lung Cancer patients: All patients with lung cancer that referred to a tertiary Oncology Unit.

SUMMARY:
In the light of a new era in the management of lung cancer this non-interventional study intend to capture all the epidemiological, clinical, pathological, molecular and treatment parameters of non-small cell (NSCLC) and small cell (SCLC) lung cancer patients from a tertiary Oncology Clinic in an Electronic Data Base (EDB).

DETAILED DESCRIPTION:
Investigators intend to build an electronic database which will record the epidemiological, clinical, pathological, molecular data and treatment parameters of lung cancer patients (NSCLC and SCLC) who are referred to a tertiary Oncology Clinic. Documentation will include: a) Patient demographics, co- morbidities, tobacco exposure in pack-years, b) Disease related parameters: method of diagnosis, histological type, disease staging (according to 7th edition of TNM for lung cancer) and metastatic sites if any, c) Molecular status: mutation status for Epidermal Growth Factor Receptor (EGFR), Anaplastic Lymphoma Kinase (ALK), Proto-oncogene tyrosine-protein kinase ROS, Hepatocyte Growth Factor Receptor (HGFRor cMET), Human Epidermal Growth Factor Receptor 2 (HER2), proto-oncogene B-Raf, and Programmed-Death Ligand 1 (PD-L1) testing when available, d) Type of treatment (surgery, radiotherapy, chemotherapy, targeted therapies, immune-therapy), and Line of treatment (neo-adjuvant, adjuvant, 1st, 2nd, 3rd, palliation therapy), e) Clinical outcome: Overall Survival (OS), Response Rate (RR), and Progression Free Survival (PFS).

ELIGIBILITY:
Inclusion Criteria:

- Since this will be a non-interventional study all adult patients who will be consent for registration of their data to EDB will be enrolled.

Exclusion Criteria:

* Patients with insufficient epidemiological or clinical data will be excluded such as patients with no demographic data or patients that have not taken at least 2 cycles of therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with lung cancer that they have been referred to our Unit will be captured to this electronic database
Sampling Method: Non-Probability Sample
Enrollment: 650 (Actual)
Dates: Start 2017-08-08 (Actual); Primary Completion 2018-12-27 (Actual); Study Completion 2018-12-27 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | 12months
  Overall Survival (OS) will be recorded for all patients and it is defined as the time in months, from diagnosis till death by any cause.

SECONDARY OUTCOMES:
Response Rate | 12 months
  Response Rate (RR) is defined as clinical or objective (imaging) response to treatment. Assessments of objective response will be done according to RECIST 1.1.All relevant data (clinical and radiological assessment) will be recorded and reported chronologically and will be correlated with the line and regimen of treatment.
Progression Free Survival | 12 months
  Progression Free Survival (PFS) will be captured for all patients. PFS is defined as the time in months, from the start of the treatment till radiological or clinical progression of the disease or death. PFS will be measured for every line of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos N Syrigos, MD,PhD, Principal Investigator — Non-Governmental, Non-Profit Organization
Locations (1):
- OCEBER, Athens, Greece